CLINICAL TRIAL: NCT01550666
Title: Treatment Development Targeting Severe and Persistent Negative Symptoms
Acronym: MOVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Dawn Velligan, Professor/Clinical Psychiatry, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HSC20110149H; R34MH093483-01 (NIH)
Record Dates: First submitted 2012-02-15; First posted 2012-03-12 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Schizophrenia
Keywords: negative symptoms
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MOVE (Experimental): MOVE Program group: MOVE consists of medication follow-up at the CHCS or ATCMHMR and meeting once a week for 9 months with a MOVE trainer in your home. You and your trainer will work on interviews for the first three visits that will talk about negative symptoms, thoughts, attitudes, and social skills that will help each of you develop goals together. Activities will be developed around improving initiation, enjoyment, success and outcome. These activities will be customized to you and will change based on your needs weekly throughout the 9 months
  Interventions: Behavioral: MOVE
- Treatment As Usual (No Intervention): Participants of this group will continue to receive medication follow up at the Center for Health Care Services. They will not be required to do anything additional except to complete assessment visits.

INTERVENTIONS:
Behavioral: MOVE — MOVE Program group: MOVE consists of medication follow-up at the CHCS or ATCMHMR and meeting once a week for 9 months with a MOVE trainer in your home. You and your trainer will work on interviews for the first three visits that will talk about negative symptoms, thoughts, attitudes, and social skills that will help each of you develop goals together. Activities will be developed around improving initiation, enjoyment, success and outcome. These activities will be customized to you and will change based on your needs weekly throughout the 9 months
  Arms: MOVE

SUMMARY:
People with schizophrenia often have problems with negative symptoms; expressing and identifying their emotions, their amount of speech, motivation and interests, feelings of purpose, social skills, and experiencing enjoyment. For this reason, new interventions are being developed to treat these problems. One new intervention is the Motivation and Engagement (MOVE) Program. The MOVE program is a new program which consists of weekly meetings for 9 months between a patient and a trainer. The weekly meetings will consist of goal setting and organization of the home to make daily tasks more manageable. During the weekly meetings the patient and trainer will discuss emotions and the trainer will help the patient identify their emotions.

The researchers hope to learn whether MOVE will help improve the problems. If it works the researchers will do a larger study comparing MOVE to other treatments that have addressed some of the problems already.

The therapist will ask you if the sessions can be audio taped to ensure that the therapist is doing a helpful job for you. They will also ask if the session can be video taped so that the tapes can be used to train other therapists learning about MOVE. The choice to do either of these is voluntary and you can continue to participate in the study if you choose not to have the session be audio and/or video taped.You will be provided a University Release document to provide that permission if you so choose.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between the 18-60 who meet DSM-IV criteria for schizophrenia confirmed by the Structured Clinical Interview Diagnosis (SCID-P version). Outpatient status.
2. Receiving treatment with antipsychotic medication
3. Clinically stable for a minimum of 5 months prior to screening (no significant changes in schizophrenia symptomatology, depressive symptoms, or community functioning, no hospitalizations, emergency visits or incarceration due to symptoms of schizophrenia or depression, no medication increases due to symptom exacerbation)
4. Has clinically meaningful negative symptoms as indicted by a score of 4 or higher on at least 2 of 6 of the following symptom domains as rated by the NSA-16; restricted affect, diminished emotional range, poverty of speech, curbing of interest, diminished sense of purpose, and diminished social drive
5. No more than moderate positive symptoms as indicated by a score of 5 or lower on BPRS-E items measuring delusions and hallucinations and no more than a 4 or higher on conceptual disorganization
6. No more than mild depression as indicated by a score of 3 or lower on the BPRS
7. No significant movement disorder as indicated by a score of 3 or lower on the ESRS-A
8. Able to provide evidence of a stable living environment (individual apartment, family home, board and care facility with no plans to move in the next year)

Exclusion Criteria:

1. History of significant head trauma
2. History of a seizure disorder
3. Mental Retardation
4. Alcohol or drug abuse or dependence within the past 3 months
5. History of violence in the past one year

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2011-01; Primary Completion 2014-08 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Changes in Negative Symptoms | 9 months after treatment
  During these times an assessor will ask questions regarding negative symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Dawn I Velligan, Ph.D., Principal Investigator — The UT Health Science Center at San Antonio
Locations (1):
- The Center for Health Care Services, San Antonio, Texas, United States